CLINICAL TRIAL: NCT01168206
Title: Assessment of Quality of Life and the Toxicity of Chemotherapy in Patients With Malignancies in Clinical Stages III and IV Under Palliative Treatment With Chemotherapy or Hormone Therapy With or Without Nutritional Supplement TK3
Brief Title: Evaluation of TK3 in Improving Quality of Life in Patients With Malignancy Under Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lavilabor Natural Products Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TK3a_FIII_Janeiro/2010
Record Dates: First submitted 2010-07-19; First posted 2010-07-23 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: 1 capsule, 3 times per day
- TK3 (Experimental): 1 capsule, 3 times per day.
  Interventions: Dietary Supplement: TK3

INTERVENTIONS:
Dietary Supplement: TK3 — Tritofano 160mg / Timina140mg and starch 150 mg
  Arms: TK3
Dietary Supplement: 1 capsule, 3 times per day — Placebo
  Arms: Placebo

SUMMARY:
The association of nutritional supplement TK3 to conventional treatment of cancer patients reduces the intensity and frequency of toxic effects and side effects caused by adjuvant or palliative treatments for the protection of healthy tissues, resulting in a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient Consent: Informed Consent and informed consent signed and dated by the patient (or his legal representative) and the professional who has obtained the consent. Must be delivered before inclusion. This term must be read and explained to the patient.
* Patients female or male, regardless of race or color.Able to ingest oral medication.
* Patients 30-80 years, with malignancy, clinical stage III or IV on chemo or hormone therapy.
* Patients who have a Karnofsky level between 60 and 80.

Exclusion Criteria:

* no agreement to sign the Deed of Consent.
* Need for use of parenteral nutrition.
* The need for food supplement already approved.
* Inability to receive the drug orally.
* Participation in another clinical trial involving chemotherapy drugs.
* Women being sexually active, which does not agree to adhere to the contraceptive methods adopted.
* Women lactating
* Any problem or condition that the investigator in the trial could be harmful to the patient.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of Quality of Life | 0 day
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 30 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 60 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 90 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 120 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 150 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.
Assessment of Quality of Life | 180 days
  Using data from the toxicity of chemotherapy and tolerability of TK3 through the clinical course of patients with malignant CS III and IV with adjuvant or palliative chemotherapy or hormone therapy, associated or not to TK3.

SECONDARY OUTCOMES:
Performance status | 0 day
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Perfomance status | 30 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Performance Status | 60 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Performance Status | 90 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Performance Status | 120 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Performance Status | 150 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Performance Status | 180 days
  Karnofsky index assesses the general condition of the patient according to the level of physical performance of the patient, which assesses the degree of functional impairment by questionnaire
Tumor Markers | 0 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 30 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 60 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 90 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 120 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 150 day
  Analysis of tumor markers specific to each tumor
Tumor Markers | 180 day
  Analysis of tumor markers specific to each tumor

CONTACTS AND LOCATIONS:
Overall Officials: Nilson Bruno Evangelista, Doctor, Principal Investigator — Lavilabor Natural Products Ltd
Locations (1):
- Sana Casa de Avaré, Avaré, São Paulo, Brazil